CLINICAL TRIAL: NCT04679025
Title: Quality Gaps in Screening and Monitoring for Postoperative Hyperglycemia in a Canadian Hospital: A Cross-sectional, Exploratory Study
Brief Title: Quality Gaps in Screening and Monitoring for Postoperative Hyperglycemia in a Canadian Hospital
Status: Completed | Type: Observational
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Shannon Ruzycki, Clinical Assistant Professor, University of Calgary
Other Study IDs: HREBA.CC-19-0157
Record Dates: First submitted 2020-12-11; First posted 2020-12-22 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: Diabetes Mellitus; Surgery; Hyperglycemia
MeSH Terms: conditions — Diabetes Mellitus; Hyperglycemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Diabetes with postoperative hyperglycemia: Patients with known diabetes (Discharge Abstract Database or hemoglobin A1c > 6.5%) who had postoperative hyperglycemia (point of care test > 10.0 mmol/L).
  Interventions: Other: Exposure - postoperative hyperglycemia
- Diabetes without postoperative hyperglycemia: Patients with known diabetes (Discharge Abstract Database or hemoglobin A1c > 6.5%) who did not have postoperative hyperglycemia (point of care test > 10.0 mmol/L).
- No diabetes with postoperative hyperglycemia: Patients without known diabetes (Discharge Abstract Database or hemoglobin A1c > 6.5%) who had postoperative hyperglycemia (point of care test > 10.0 mmol/L).
  Interventions: Other: Exposure - postoperative hyperglycemia
- No diabetes and no postoperative hyperglycemia: Patients without known diabetes (Discharge Abstract Database or hemoglobin A1c > 6.5%) who did not have postoperative hyperglycemia (point of care test > 10.0 mmol/L).

INTERVENTIONS:
Other: Exposure - postoperative hyperglycemia — Postoperative hyperglycemia (blood or capillary glucose > 10.0 mmol/L) within 72 hours of a surgical procedure
  Groups: Diabetes with postoperative hyperglycemia; No diabetes with postoperative hyperglycemia

SUMMARY:
Patients with and without diabetes who have postoperative hyperglycemia have worse outcomes than patients with in-target blood sugars. Previous quality improvement work suggests numerous barriers and clinical inertia may contribute to quality gaps in glycemic management for surgical patients. Using a framework for perioperative glycemic management, we sought to measure quality gaps in perioperative glycemic care.

This cross-sectional study used administrative data to measure the proportion of surgical patients with and without known diabetes who underwent preoperative hemoglobin A1c measurement, postoperative point-of-care testing for glucose (POCT), had hyperglycemia, and received basal bolus insulin regimens for treatment. We performed an exploratory analysis comparing length of stay (LOS) in patients with and without diabetes who had and did not have postoperative hyperglycemia.

ELIGIBILITY:
Inclusion Criteria:

* Underwent inpatient surgical procedure at the Foothills Medical Centre between Apr 1 2019 and March 31 2020
* Stayed in hospital for more than 24-hours after surgery

Exclusion Criteria:

* Younger than 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients undergoing a surgical procedure at the Foothills Medical Centre who were admitted for at least 24-hours.
Sampling Method: Non-Probability Sample
Enrollment: 7633 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Number of point of care blood glucose measurements in 24-hours after surgery | 24-hours post surgery
Proportion of patients who have hyperglycemia | 24-hours after surgery
  blood or capillary glucose > 10 mmol/L

SECONDARY OUTCOMES:
Proportion of patients who have moderate hyperglycemia | 24-hours after surgery
  blood or capillary glucose 14.0-17.9 mmol/L
Proportion of patients who have severe hyperglycemia | 24-hours after surgery
  blood or capillary glucose > 18.0 mmol/L
Hospital Length of stay | Until study completion (up to one year from surgical procedure)
  Hospital length of stay (days)

CONTACTS AND LOCATIONS:
Locations (1):
- Foothills Medical Centre, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Yes
Data is available from the study principal investigator upon reasonable request.
Supporting Information: Study Protocol, SAP
Time Frame: Present for five years after study completion (March 31 2020).
Access Criteria: Email shannon.ruzycki@ucalgary.ca